CLINICAL TRIAL: NCT03267043
Title: Family Nurture Intervention in the NICU at The Valley Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G Welch, Associate Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology), Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: AAAR4899
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Premature Birth; Obstetric Labor, Premature
Keywords: preterm birth; NICU; neonatal; skin to skin; kangaroo care; separation stress; family nurture; maternal confidence; maternal competence; calming cycle; infant neurodevelopment; infant psychological development; mother-infant co-regulation; postpartum depression
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care (Active Comparator): Participants enrolled in Phase 1 will be receiving the current standard of care in the NICU at The Valley Hospital.
  Interventions: Behavioral: Standard Care
- Family Nurture Intervention (FNI) (Experimental): Participants enrolled in Phase 2 will be receiving family nurture intervention (FNI) that focuses on supporting the parents and facilitating emotional connection between mother and infant during the infant's NICU stay.
  Interventions: Behavioral: Family Nurture Intervention (FNI)
- Standard Care - Case Studies (Active Comparator): Participants enrolled as case studies in Phase 1 will be receiving the current standard of care in the NICU at The Valley Hospital. These participants will be those who fall outside the inclusion criteria.
  Interventions: Behavioral: Standard Care
- FNI - Case Studies (Experimental): Participants enrolled in Phase 2 will be receiving family nurture intervention (FNI) that focuses on supporting the parents and facilitating emotional connection between mother and infant during the infant's NICU stay. These fall outside the inclusion criteria but act as a comparator to the case studies of Phase 1.
  Interventions: Behavioral: Family Nurture Intervention (FNI)

INTERVENTIONS:
Behavioral: Family Nurture Intervention (FNI) — Subjects will be guided by the nursing staff through an enhanced program of mother/infant interactions, which include skin-to-skin holding.
  Other Names: FNI
  Arms: FNI - Case Studies; Family Nurture Intervention (FNI)
Behavioral: Standard Care — Established routine care provided on the NICU floor by specially trained health care professionals.
  Other Names: SC
  Arms: Standard Care; Standard Care - Case Studies

SUMMARY:
The purpose of this study is to compare neurodevelopment and activity in infants born preterm (25 to 34 1/7 weeks gestational age (GA)) receiving Standard Care (SC) or Family Nurture Intervention (FNI) in the neonatal intensive care unit (NICU).

The investigators hypothesize that FNI will improve: i) neonatal electroencephalographic activity ii) maternal caregiving and wellbeing (psychological and physiological, and iii) infant behavior and neurodevelopment at 18 months corrected age (CA).

The two-phase effectiveness study aims to:

* Phase 1 - Examine the existing Standard Care Approximately 35 infants and their mothers
* Phase 2 - Examine effectiveness by implementing FNI unit-wide so that every baby receives the intervention Approximately 35 infants and their mothers

DETAILED DESCRIPTION:
This study aims to build upon the findings of the earlier randomized controlled trial (RCT) conducted at the Columbia University Medical Center (CUMC) comparing effects, both physiological and emotional, of the current standard method of encouraging contact between mothers and their babies in the NICU with the more specific approach of Family Nurture Intervention (FNI). In addition to receiving standard care, NICU families assigned to FNI received added intervention that focused on supporting the parents and facilitating emotional connection between mother and infant during the infant's NICU stay.

The investigators wish to conduct an effectiveness trial to evaluate if the family nurture intervention's findings can be replicated on a unit-wide level. This effectiveness trial will take place over two parts. There will be two groups; standard care (SC) and intervention (FNI). Phase 1 of the effectiveness study will evaluate the standard care (SC) group in the unit as a baseline measurement and point of comparison to determine if unit-wide FNI reproduces its prior findings (Phase 2). The standard care group (Phase 1) will receive the current standard of care in the NICU. In Phase 2, FNI will be implemented unit-wide, but infants born between 26 weeks and 0 days to 33 weeks 6 days gestation will be eligible to be enrolled into the study. In addition to receiving standard care, patients enrolled during phase 2 will receive added interventions from the trained FNI nursing staff. These added interventions will include supporting the parents and facilitating contact between mother and infant during their infant's NICU stay.

ELIGIBILITY:
For the Standard Care and FNI Groups

Inclusion Criteria:

* infant is between 26 and 33 6/7 weeks gestational age upon admission
* infant is a singleton or twin

Exclusion Criteria:

* infant's attending physician does not recommend enrollment in the study
* severe congenital anomalies including chromosomal anomalies
* ultrasound evidence of large parenchymal hemorrhagic infarction (>2 cm, intraventricular hemorrhage grade 3 or 4)
* infant cardiac anomalies
* mother has known history of substance abuse, severe psychiatric illness or psychosis
* status of enrolled subject changes and subject now falls into exclusion criteria
* mother and/or infant has a medical condition that precludes intervention components
* mother and/or infant has a contagion that endangers other participants in the study

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
EEG Power in the frontal polar region | Up to 41 weeks gestational age
  Measured in microvolts (µV)^2 for infants.

SECONDARY OUTCOMES:
EEG Coherence in the left frontal polar to right frontal polar region | Up to 41 weeks gestational age
  Coherence is a number between 0-1, generated by looking at the similarity/differences in activity between brain regions through analysis of EEG.
CES-D Score | Up to 18 months
  To examine maternal depression, the Center for Epidemiologic Studies Depression Scale (CES-D) is a 20 item self-report inventory designed to assess current but nonspecific distress rather than clinically diagnosed depression. It is the most frequently used measure in the field of infant research and maternal depression. Items probe for depressive symptoms and attitudes within the past week.
State-Trait Anxiety Inventory (STAI) Score | Up to 18 months
  To examine Maternal Anxiety, the State-Trait Anxiety Inventory (STAI) comprises 2 separate self-report scales of 20 items each that measure state and trait anxiety. The S-Anxiety Scale (measuring state), has been found to be a sensitive indicator of changes in transitory anxiety experienced by patients in counseling, psychotherapy, and behavior-modification programs, and has been used to assess the level of anxiety induced by unavoidable real-life stressors. The T-Anxiety scale has proven useful for identifying persons who differ in motivation or drive level. The STAI has been used in studies examining parents of hospitalized children, the transition to a maternal role, perception of illness severity in infants, and maternal anxiety during pregnancy and fetal attachment.
Neurobehavioral Assessments of Infants - Bayley Scales or Infant and Toddler Development, Bayley III | Up to 18 months
  At the 18 month corrected age follow-up, infants are administered the Bayley Scales of Infant and Toddler Development, Bayley III consisting of three developmental domains: Cognitive, Language (receptive/expressive) and Motor (fine/gross). For each domain, a composite score is provided and is scaled to a mean score of 100 and a standard deviation of 15. A child will receive 1 point for every item successfully completed. The administration of each section will end if the child received 0 points on 5 consecutive items. Scores <70 indicate significant developmental delays and scores <80 indicate mild to moderate developmental delays.
  Cognitive Scale - comprised of 91 items Language Scale - comprised of 97 items Motor Scale - comprised of 138 items

OTHER OUTCOMES:
Welch Emotional Connection Scale | Up to 18 months
  To examine Mother-Infant Emotional Connection, this is a brief 4-item assessment requiring 5 minutes or less, which assesses the character of the relationship between study mothers and infants. It is filled out by study staff who rate mothers and infants in a dyadic interaction on their attraction, their vocal communication, facial expressiveness, and sensitivity and responsivity towards each other.
Child Behavior Checklist Score | Up to 18 months
  The Child Behavior Checklist (CBCL) is a device by which parents rate their child's problem behaviors and competencies. The CBCL can also be used to measure a child's change in behavior over time or following a treatment. The CBCL consists of 100 items. This will be administered at the 18 Months CA Follow-Up.
Modified Checklist for Autism in Toddlers (M-CHAT) Score | Up to 18 months
  The M-CHAT is a questionnaire validated for screening toddlers to assess risk for autism spectrum disorders (ASD). It is a 23 yes/no item questionnaire administered to the mother which can be scored in less than 2 minutes. This will be administered at the 18 Month CA Follow-Up.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - The Valley Hospital, Ridgewood, New Jersey
  - Morgan Stanley Children's Hospital of New York (MSCHONY), New York, New York

IPD SHARING:
Plan to Share IPD: Undecided